CLINICAL TRIAL: NCT01083446
Title: A Nutritional Approach to Minimal Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof' Nachum Vaisman, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-NV-236; 0236-08-TLV
Record Dates: First submitted 2008-06-17; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2008-06

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: Encephalopathy; Cirrhotics
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Nutritional intervention, standard Israeli breakfast
  Interventions: Other: Nutritional Intervention
- B (Active Comparator): Nutritional Intervention, fast
  Interventions: Other: Nutritional Intervention

INTERVENTIONS:
Other: Nutritional Intervention — Cognitive and executive functions before and after standard israeli breakfast (30% of caloric value and 21 gram protein)
  Arms: A
Other: Nutritional Intervention — Cognitive and executive functions during fast
  Arms: B

SUMMARY:
This trial will study a possible effect of standard Israeli breakfast (30% of caloric value and 21 gram protein) on cognitive and executive functions (working memory, visual memory, concentration and coordination), on patients with mild-moderate liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* All consented adults (age > 18), with the diagnosis of CHILD A cirrhosis with MELD score of < 10.
* Diagnosis of liver cirrhosis as documented by liver biopsy (stage IV) and / or fibroscan (score > 12 kpa) and / or fibrotest (score > 0.74) and /or imaging.

Exclusion Criteria:

* History of > grade II hepatic encephalopathy (HE).
* Diagnosis of dementia, Parkinson disease, Schizophrenia (Patients with major depression will be noted but not excluded).
* Use of sedatives, tranquilizers or anti- psychotic medication during and/or 2 weeks prior to enrolling Use of antibiotics for any length of period during and/or 2 weeks prior to enrolling.
* Current use of lactulose or neomycin.
* Use of alcohol or elicit drugs during and/ or 6 months prior to enrolling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof', Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel, Israel

REFERENCES:
- [Derived] Vaisman N, Katzman H, Carmiel-Haggai M, Lusthaus M, Niv E. Breakfast improves cognitive function in cirrhotic patients with cognitive impairment. Am J Clin Nutr. 2010 Jul;92(1):137-40. doi: 10.3945/ajcn.2010.29211. Epub 2010 May 5. PMID 20444959